CLINICAL TRIAL: NCT05682183
Title: A Community-based Multi-domain Psychoeducation Self-management Programme (MPSP) for Adults With Major Depressive Disorder in Singapore : A Pilot Randomized Controlled Trial
Brief Title: Multi-domain Psychoeducation Self-management Program for Adults With MDD in Singapore
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Goh Yong-Shian, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: MPSP_2022
Record Dates: First submitted 2022-12-15; First posted 2023-01-12 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Community dwelling adults
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-domain Psychoeducation Self-management Programme (Active Comparator): Participants will be registered at the care centre and will receive usual care from their care manager who is assigned to them when they register with the centre. Those who are randomised into the intervention arm will undergo 5-sessions of Multi-domain Psychoeducation Self-management Programme over 5 weeks.
  Interventions: Behavioral: Multi-domain Psychoeducation Self-management Programme
- Treatment as Usual (Active Comparator): Participants will be registered at the care centre and will receive usual care from their care manager who is assigned to them when they register with the centre.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Multi-domain Psychoeducation Self-management Programme — The MPSP is a 5-weeks psychoeducation programme aimed at improving the biopsychosocial health of people with MDD (PMDD). It will be conducted on every Saturday in the morning, afternoon and evening. Specific time of each session will be further discussed with the centre. Each session will last for approximately 45 minutes to 60 minutes and will be capped at 10 participants. The mode of session will be face-to-face (F2F) session conducted at MindCare.
  Arms: Multi-domain Psychoeducation Self-management Programme
Other: Treatment as usual — Care management from assigned care manager
  Arms: Treatment as Usual

SUMMARY:
This is a single-centre, two-arm, unblinded pilot randomised controlled trial study on 60 participants (30 in each arm) from the community mental health service (CMHS) centre within a social service agency in Singapore based on inclusion criteria. The study will examine the effects of a 5-sessions of Multi-domain Psychoeducation Self-management Programme and treatment-as-usual) over 5 weeks or control (treatment-as-usual) group.

DETAILED DESCRIPTION:
This is a single-centre, two-arm, unblinded pilot randomised controlled trial study. A total of 60 participants (30 in each arm) will be conveniently recruited from the community mental health service (CMHS) centre within a social service agency in Singapore based on inclusion criteria. Block randomisation with a block size of two will be used to randomise participants into the intervention (5-sessions of Multi-domain Psychoeducation Self-management Programme and treatment-as-usual) over 5 weeks or control (treatment-as-usual) group. Primary outcomes measures which include self-management competence, self-efficacy to manage emotions, mental health quality of life and depressive symptoms severity, will be collected at three timepoints: (T1) baseline, (T2) immediately post-intervention and (T3) three months post-intervention. Quantitative data will be analysed using the Statistical Package for Social Sciences (SPSS) software using non-parametric tests. Secondary outcomes include the feasibility and acceptability of the MPSP. Feasibility of the intervention will be evaluated using pre-defined recruitment, attendance and follow-up rates. Acceptability of the intervention will be evaluated using a semi-structured interview guide based on the Theoretical Framework of Acceptability, immediately post-intervention (T2) or not more than a week from the last session. Data for acceptability will be transcribed verbatim and thematically analysed based on Braun and Clarke's thematic analysis guideline.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with Major Depressive Disorder
* Community-dwelling adults aged 21 to 80 years old
* Singaporean or permanent residents
* Literate in the English language
* Willing to be video or audio-recorded during the qualitative interview sessions for acceptability of intervention

Exclusion Criteria:

* Clinically diagnosed with maternal depression
* Clinically diagnosed with cognitive impairment/ intellectual disability
* Pregnant women
* Currently institutionalised in a long-term care facility
* Currently attending other psychoeducation self-management programmes
* Those who do not agree to the audio or video recording.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Management Self-Test (T1) | (T1) baseline (before the start of intervention)
  The self-reported 5-item scale measures the degree of perceived competence of self-management among individuals with or without psychiatric disorders. Each item consists of a 5-point Likert scale, with a score of '0' indicating poor self-management and '4' excellent self-management; hence, higher score represents better perceived self-management practice. The lowest possible score for this scale is 0 and the highest possible score for the scale is 25.
Self-Management Self-Test (T2) | (T2) directly post-intervention (on the day of the final session)
  The self-reported 5-item scale measures the degree of perceived competence of self-management among individuals with or without psychiatric disorders. Each item consists of a 5-point Likert scale, with a score of '0' indicating poor self-management and '4' excellent self-management; hence, higher score represents better perceived self-management practice. The lowest possible score for this scale is 0 and the highest possible score for the scale is 25.
Self-Management Self-Test (T3) | (T3) three months post-intervention.
  The self-reported 5-item scale measures the degree of perceived competence of self-management among individuals with or without psychiatric disorders. Each item consists of a 5-point Likert scale, with a score of '0' indicating poor self-management and '4' excellent self-management; hence, higher score represents better perceived self-management practice. The lowest possible score for this scale is 0 and the highest possible score for the scale is 25.
Patient Reported Outcomes Measurement Information System (PROMIS) Self-efficacy for Managing Chronic Conditions- Managing Emotions (T1) | (T1) baseline (before the start of intervention)
  The self-reported 8-item scale specifically evaluates an individual's confidence to manage or control symptoms of anxiety, depression, helplessness and discouragements, amongst others. Each item consists of a 5-point Likert scale, with a score of' 1' indicating the least confidence and '5' indicating the utmost confidence; hence, a higher score represents greater self-efficacy. The lowest possible score for this scale is 8 and the highest possible score for the scale is 40.
Patient Reported Outcomes Measurement Information System (PROMIS) Self-efficacy for Managing Chronic Conditions- Managing Emotions (T2) | (T2) directly post-intervention (on the day of the final session)
  The self-reported 8-item scale specifically evaluates an individual's confidence to manage or control symptoms of anxiety, depression, helplessness and discouragements, amongst others. Each item consists of a 5-point Likert scale, with a score of' 1' indicating the least confidence and '5' indicating the utmost confidence; hence, a higher score represents greater self-efficacy. The lowest possible score for this scale is 8 and the highest possible score for the scale is 40.
Patient Reported Outcomes Measurement Information System (PROMIS) Self-efficacy for Managing Chronic Conditions- Managing Emotions (T3) | (T3) three months post-intervention.
  The self-reported 8-item scale specifically evaluates an individual's confidence to manage or control symptoms of anxiety, depression, helplessness and discouragements, amongst others. Each item consists of a 5-point Likert scale, with a score of' 1' indicating the least confidence and '5' indicating the utmost confidence; hence, a higher score represents greater self-efficacy. The lowest possible score for this scale is 8 and the highest possible score for the scale is 40.
Mental Health Quality of Life Questionnaire (T1) | (T1) baseline (before the start of intervention)
  The self-administered 7-item scale measures the quality of life of an individual based on the context of mental health. It was developed based on seven quality of life dimensions: self-image; independence; mood; relationships; daily activities; physical health and; future. Each item has a 4-point response level. An overall index score will be calculated based on the summation of each item's score; higher scores indicate better quality of life. The lowest possible score for this scale is 7 and the highest possible score for the scale is 28.
Mental Health Quality of Life Questionnaire (T2) | (T2) directly post-intervention (on the day of the final session)
  The self-administered 7-item scale measures the quality of life of an individual based on the context of mental health. It was developed based on seven quality of life dimensions: self-image; independence; mood; relationships; daily activities; physical health and; future. Each item has a 4-point response level. An overall index score will be calculated based on the summation of each item's score; higher scores indicate better quality of life. The lowest possible score for this scale is 7 and the highest possible score for the scale is 28.
Mental Health Quality of Life Questionnaire (T3) | (T3) three months post-intervention.
  The self-administered 7-item scale measures the quality of life of an individual based on the context of mental health. It was developed based on seven quality of life dimensions: self-image; independence; mood; relationships; daily activities; physical health and; future. Each item has a 4-point response level. An overall index score will be calculated based on the summation of each item's score; higher scores indicate better quality of life. The lowest possible score for this scale is 7 and the highest possible score for the scale is 28.
Patient Health Questionnaire (PHQ-9) (T1) | (T1) baseline (before the start of intervention)
  The self-reported 9-item scale is a dual-purpose scale that measures the severity of depressive symptoms. All items have a 4-point Likert scale, with '0' indicating 'not at all' and '3' indicating 'nearly every day'; higher scores represent greater severity of depression. The summation of scores can be categorised to represent depression severity: 0-4 indicates none to minimal severity; 5-9 indicates mild severity; 10-14 indicates moderate severity; 15-19 indicates moderately severe and; 20-27 indicates severe depression (PHQ Screeners, 2002).
Patient Health Questionnaire (PHQ-9) (T2) | (T2) directly post-intervention (on the day of the final session)
  The self-reported 9-item scale is a dual-purpose scale that measures the severity of depressive symptoms. All items have a 4-point Likert scale, with '0' indicating 'not at all' and '3' indicating 'nearly every day'; higher scores represent greater severity of depression. The summation of scores can be categorised to represent depression severity: 0-4 indicates none to minimal severity; 5-9 indicates mild severity; 10-14 indicates moderate severity; 15-19 indicates moderately severe and; 20-27 indicates severe depression (PHQ Screeners, 2002).
Patient Health Questionnaire (PHQ-9) (T3) | (T3) three months post-intervention.
  The self-reported 9-item scale is a dual-purpose scale that measures the severity of depressive symptoms. All items have a 4-point Likert scale, with '0' indicating 'not at all' and '3' indicating 'nearly every day'; higher scores represent greater severity of depression. The summation of scores can be categorised to represent depression severity: 0-4 indicates none to minimal severity; 5-9 indicates mild severity; 10-14 indicates moderate severity; 15-19 indicates moderately severe and; 20-27 indicates severe depression (PHQ Screeners, 2002).

CONTACTS AND LOCATIONS:
Locations (1):
- Alice Lee Centre for Nursing Studies, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No